CLINICAL TRIAL: NCT02748902
Title: An Open Label Exploratory Study Evaluating the Efficacy and Safety of Ingenol Mebutate 0.05% Gel for the Treatment of Verruca Vulgaris.
Brief Title: Exploratory Study of Efficacy and Safety of Ingenol Mebutate 0.05% Gel for Common Warts on the Hands.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neal D. Bhatia, MD (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor-Investigator, Neal D. Bhatia, MD, Director, Clinical Dermatology, TCR Medical Corporation
Organization: TCR Medical Corporation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCR-202i-03-16
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Verruca Vulgaris; Common Warts
Keywords: Verruca vulgaris; Common warts; Verruca; Warts; Papilloma virus; ingenol mebutate 0.05% gel; hands
MeSH Terms: conditions — Warts | interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ingenol mebutate 0.05% gel (Experimental): Single group, open label. All subjects will receive active product.
  Interventions: Drug: ingenol mebutate 0.05% gel

INTERVENTIONS:
Drug: ingenol mebutate 0.05% gel — Ingenol mebutate 0.05% gel applied to a minimum of two and a maximum of five common warts on days 1 and 2.
  Other Names: Picato®

SUMMARY:
The purpose of this study is to determine if ingenol mebutate 0.05% gel is safe and effective in treating common warts on the hands.

DETAILED DESCRIPTION:
This is an open label exploratory study evaluating the efficacy and safety of ingenol mebutate 0.05% gel for the treatment of verruca vulgaris. The study will be conducted at one site with one investigator, all subjects will receive active drug. Prior to the application of the investigational product (IP) on Day 1, the individual warts will be pared down with a 15 blade up to obtain debridement of intact skin to maximize exposure and allow for effective penetration of therapy into the lesion.

Subjects can be screened for the study up to 45 days before Visit 1. During screening, the study requirements will be reviewed, written informed consent obtained, and eligibility confirmed. If applicable, qualified subjects can washout from prohibited medications or treatments prior to Visit 1 once they have been consented. These procedures may be combined with Visit 1.

There will be one treatment arm, all subjects receive active ingenol mebutate 0.05% gel once daily for two consecutive days to lesions. Each subject will be screened for inclusion. The treatment will be applied to the entire wart lesion(s) and 0.5 cm margin around the lesion(s). All treatments will be applied in the clinic. A minimum of two (2) and a maximum of five (5) warts will be treated. In addition, one of the two warts will be identified for treatment with occlusion with a bandage each day for 24 hours after each application.

The subjects will be evaluated at Day 1 and Day 2 when the consecutive applications of investigational product will be applied, then at Day 8, 29 and 57 to evaluate anticipated efficacy outcomes (lesion size, clearance, etc.) as well as assess for adverse events/SAEs. The wart that is identified for occlusion will be treated with investigational product and occluded for 24 hours after each application of IP. Subjects will be instructed to avoid excessive exposures to water or other potential contactants or irritants after application of the IP for the following 48 hours to avoid transfer of the IP.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female 18 years of age or older. Females must be post-menopausal, surgically sterile, or using a medically acceptable form of birth control with a negative urine pregnancy test at Visit 1. For the purpose of this study, the following are considered medically acceptable methods of birth control: Oral Contraceptives, Contraceptive patches, Contraceptive Injection (Depo-Provera®), Contraceptive Implant (Implanon™), Essure®, Vaginal Contraceptive (Nuva-Ring®), IUD, hormonal IUD (Mirena®); double-barrier methods (e.g. condom and spermicide), sterile partner (e.g., vasectomy performed at least six months prior to the subject's initiation of treatment) and abstinence with a documented second acceptable method of birth control should subject become sexually active.
2. Subject has provided written informed consent.
3. Subject has at least two (2) verrucous papules diagnosed as common wart (verruca vulgaris) by the investigator on the hands excluding proximity to the nails (periungual warts) at Visit 1.
4. Subject is willing and able to have the investigational product (IP) applied at Visits 1 and 2, comply with study instructions and commit to all follow-up visits for the duration of the study.
5. Subject is in good general health and free of any disease state or physical condition that might impair evaluation of wart lesions or which, in the investigator's opinion, exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject is currently enrolled in an investigational drug or device study.
3. Subject has used an investigational drug or investigational device treatment within 30 days prior to the Visit 1.
4. Subject has a history of prior treatment with ingenol mebutate gel.
5. Subject is immunosuppressed (HIV, organ transplant, systemic malignancy, etc.) in the opinion of the investigator.
6. Subject has a history of injury to lesions or treatment area in the past 30 days.
7. Subject has a history of sensitivity to any of the ingredients in the investigational product.
8. Subject used any topical agents (including dry powder, bland emollients, non-medicated lotions, etc.) within a 3 cm border of the area to be treated within 14 days prior to entry into the study.
9. Subject has used topical medications such as corticosteroids, alpha-hydroxyacids greater than 5% (e.g., glycolic acid, lactic acid, etc.), beta-hydroxyacids greater than 2% (e.g., salicylic acid), urea greater than 5%, or topical retinoids (e.g., tazarotene, adapalene, tretinoin) adjacent to or within a 3 cm border around the area to be treated within 28 days prior to entry into the study.
10. Subject has used cryotherapy to lesions adjacent to or within a 3 cm border around the area to be treated within 2 weeks prior to entry into the study.
11. Subject has used systemic steroid therapy (e.g., methylprednisolone, predinisone) or NSAIDs within 7 days from Visit 1/Day 1 or initiation during the study. *Subjects may use Tylenol (Acetaminophen) for pain relief, as needed, throughout the study. Subjects may use low dose aspirin (81mg) for cardiac prophylaxis throughout the study.*
12. Subject has used chemotherapeutic agents, immunosuppressive agents, or retinoids within 4 weeks prior to entry into the study.
13. Subject has applied topical treatment such as 5-FU, imiquimod, diclofenac sodium, sinecatechins ointment, or other treatments either indicated or off-label for warts to lesions adjacent to (within a 3 cm border around the Treatment Area) or within the selected Treatment Area within 90 days prior to entry into the study.
14. Subject has had any prior intralesional treatment of the warts including injection of candida antigen, 5-FU, and bleomycin.
15. Subject has any condition in the Treatment Area that would impact the treatment or proper assessment of the outcome (e.g. scarring, marked dermatitis, etc.) in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Efficacy assessed by verruca vulgaris lesion counts (total number of lesions present) | Day 1 through Day 57
  Total number of warts in the treatment area will be counted and assessed for clearance

SECONDARY OUTCOMES:
Safety assessed by number and severity of adverse events reported | Day 1 through Day 57
  All adverse events that occur during the study (from the time of informed consent) will be recorded.
Safety assessed by application site reactions on a 5 point scale (0/clear - 4/severe) | Day 1 through Day 57
  Application site reactions defined as of erythema, flaking/scaling, crusting, swelling, erosion/ulceration and vesiculation/pustulation.

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Bhatia, MD, Principal Investigator — TCR Medical Corporation
Locations (1):
- Therapeutics Clinical Research, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data will be collected and reported in aggregate through peer reviewed journal publication and/or poster presentations.

REFERENCES:
- [Background] Lebwohl M, Swanson N, Anderson LL, Melgaard A, Xu Z, Berman B. Ingenol mebutate gel for actinic keratosis. N Engl J Med. 2012 Mar 15;366(11):1010-9. doi: 10.1056/NEJMoa1111170. PMID 22417254
- [Background] Schopf RE. Ingenol mebutate gel is effective against anogenital warts - a case series in 17 patients. J Eur Acad Dermatol Venereol. 2016 Jun;30(6):1041-3. doi: 10.1111/jdv.13097. Epub 2015 Mar 28. No abstract available. PMID 25820019